CLINICAL TRIAL: NCT04742907
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 2 Trial to Evaluate the Safety and Efficacy of TU-100 as an Adjunct to an Enhanced Recovery After Surgery (ERAS) Protocol in Subjects Undergoing Bowel Resection
Brief Title: Safety and Efficacy of TU-100 as an Adjunct to an Enhanced Recovery After Surgery in Subjects Undergoing Bowel Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tsumura USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TU100P2T4
Record Dates: First submitted 2021-01-29; First posted 2021-02-08 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Enhanced Recovery After Surgery
MeSH Terms: interventions — 12,13-dihydro-N-methyl-6,11,13-trioxo-5H-benzo(4,5)cyclohepta(1,2-b)naphthalen-5,12-imine; dai-kenchu-to

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Investigator
Masking Description: Investigators, study staff, sponsor designees, and subjects will be blinded to randomized study treatment for the duration of the study. The pharmacist or designee performing the preparation and administration will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TU-100 15 g/day (Experimental): Subjects will receive a total daily dose of TU-100 5 g TID until hospital discharge or ≤ 10 days (whichever is earlier).
  Interventions: Drug: TU-100
- TU-100 7.5 g/day (Experimental): Subjects will receive a total daily dose of TU-100 2.5 g TID until hospital discharge or ≤ 10 days (whichever is earlier).
  Interventions: Drug: TU-100
- Placebo (Placebo Comparator): Subjects will receive placebo TID until hospital discharge or ≤ 10 days (whichever is earlier).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TU-100 — Treatment with investigational product
  Other Names: Daikenchuto
  Arms: TU-100 15 g/day; TU-100 7.5 g/day
Drug: Placebo — Treatment with placebo product
  Arms: Placebo

SUMMARY:
This multicenter, randomized, double-blinded, placebo-controlled study will evaluate the effect of TU-100 on resolution of postoperative ileus (POI) in subjects undergoing open or laparoscopic bowel resection (BR).

DETAILED DESCRIPTION:
Subjects will be screened up to 28 days before their planned surgery and will be randomized 1:1:1 (TU-100 15 g/day: TU-100 7.5 g/day: placebo) on postoperative Day 1 before the first dose of study medication. After randomization, subjects will receive a total daily dose of TU-100 15g, TU-100 7.5 g, or matching placebo (3 times per day (TID)) until hospital discharge or ≤ 10 days (whichever is earlier). All subjects will be treated with study medication as adjunct to an enhanced recovery (ERAS) pathway for gastrointestinal (GI) recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Women of childbearing potential (WOCBP) or men whose sexual partners are WOCBP; must be able and willing to use at least 1 highly effective method of contraception during the study and for 30 days after the last dose of study drug
3. American Society of Anesthesiologists Physical Status Score of 1 to 3
4. Scheduled for an elective BR via open or laparoscopic approach
5. Ability to understand the study procedures, have agreed to participate in the study program, and have voluntarily provided informed consent

Exclusion Criteria:

1. Scheduled for a BR that is not listed in this protocol
2. Requires any additional resections beyond the intestine (eg, hepatectomy, distal pancreatectomy, pancreaticoduodenectomy, gastric resection, uterine resection), or concomitant surgeries (with the exception of biopsies)
3. Requires the formation of a stoma (ileostomy or colostomy)
4. History of surgeries, illness, or behavior (eg, depression, psychosis) that in the opinion of the investigator might confound the study results or pose additional risk in administering the study procedures
5. Have a functional colostomy or ileostomy
6. Diagnosed with advanced or metastatic colon cancer (Stage IV by tumor, node, and metastasis classification)
7. Positive coronavirus disease 2019 (COVID-19) test
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (including human immunodeficiency virus (HIV)), diabetes, symptomatic congestive heart failure and ejection fraction < 35%, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with protocol requirements
9. Chronic pain syndrome unrelated to the planned surgery requiring consistent management with analgesics and/or other non-pharmacologic modalities
10. Myocardial infarction within 3 months
11. Corrected QT interval > 500 msec
12. Diabetic gastroparesis
13. Compromised immune system, either from treatment with corticosteroids or other immunosuppressive agent within 2 weeks of surgery or from immunosuppressive disease (HIV)
14. Pregnant (identified by a positive serum pregnancy test) or lactating, or are not postmenopausal (no menses for at least 1 year) and are of childbearing potential and not using an accepted method of birth control (surgical sterilization, intrauterine contraceptive device, oral contraceptive, diaphragm, or condom in combination with contraceptive cream, jelly, or foam or abstinence)
15. Participated in another investigational drug/biologic or medical device study within 30 days of surgery or will be enrolled in another investigational drug or medical device study, or any study in which active subject participation is required outside routine hospital data collection during the course of the study
16. Illicit drug use or alcohol abuse based on medical history, or currently engaged in illicit drug use or alcohol abuse
17. Uses of supplemental ginger, ginseng, or Zanthoxylum fruit within 72 hours before randomization
18. Has a history of allergic reactions to ginseng, ginger, Zanthoxylum fruit, or lactose
19. Has clinical symptoms of lactose intolerance after ingesting milk or milk-containing products (abdominal pain, flatulence, diarrhea)
20. Unwilling or unable to comply with procedures described in this protocol or is otherwise unacceptable for enrollment in the opinion of the investigator
21. Has a history of previous surgeries, illness (interstitial pneumonia), or behavior (depression, psychosis) that, in the opinion of the investigator, might confound the study results or pose additional risk in administering the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Florence Site, Florence, Alabama
  - Gilbert Site, Gilbert, Arizona
  - Little Rock Site, Little Rock, Arkansas
  - Duarte Site, Duarte, California
  - Los Angeles Site #1, Los Angeles, California
  - Los Angeles Site #2, Los Angeles, California
  - Palo Alto Site, Palo Alto, California
  - Sacramento Site, Sacramento, California
  - Danbury Site, Danbury, Connecticut
  - Clearwater Site, Clearwater, Florida
  - Orlando Site, Orlando, Florida
  - Tampa Site, Tampa, Florida
  - Weston Site, Weston, Florida
  - Chicago Site #2, Chicago, Illinois
  - Chicago Site #1, Chicago, Illinois
  - Urbana Site, Urbana, Illinois
  - Lexington Site, Lexington, Kentucky
  - Metairie Site, Metairie, Louisiana
  - Boston Site #1, Boston, Massachusetts
  - Detroit Site, Detroit, Michigan
  - St. Louis Site, St Louis, Missouri
  - Newark Site, Newark, New Jersey
  - Mineola Site, Mineola, New York
  - New York Site, New York, New York
  - Stony Brook Site, Stony Brook, New York
  - Cleveland Site #2, Cleveland, Ohio
  - Cleveland Site #1, Cleveland, Ohio
  - Philadelphia Site #2, Philadelphia, Pennsylvania
  - Pittsburgh Site, Pittsburgh, Pennsylvania
  - Charleston Site, Charleston, South Carolina
  - Memphis Site, Memphis, Tennessee
  - Dallas Site, Dallas, Texas
  - Fort Worth Site, Fort Worth, Texas
  - Salt Lake City Site, Salt Lake City, Utah
  - Roanoke Site, Roanoke, Virginia
  - Milwaukee Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Nedeljkovic SS, Silinsky JD, Nagle D, Lee SW, Ayad S, Segura-Vasi AM, Fleshner PR, Choti MA, Wren SM, Kosaka B Pharm J, Tanaka Y, Li YP, Rachfal AW, Techner LM, Gan TJ, Fichera A, Michelassi F. Evaluation of TU-100 (Daikenchuto), a Traditional Japanese Kampo Medicine, as an Adjunct to Enhanced Recovery After Surgery, for Acceleration of Gastrointestinal Recovery After Bowel Resection: Results of a Proof-of-Concept, Phase 2, Randomized, Double-Blinded, Placebo-Controlled Trial. Dis Colon Rectum. 2026 Jan 1;69(1):73-86. doi: 10.1097/DCR.0000000000003990. Epub 2025 Oct 20. PMID 41114550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was carried out at 36 sites in the United States (US).
Period: Overall Study
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo
Started | 134 | 134 | 134
Safety (Baseline) Analysis Set | 132 | 130 | 130
Completed | 120 | 114 | 120
Not Completed | 14 | 20 | 14
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Lost to Follow-up | 3 | 3 | 2
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 6 | 4
Not completed — Subject Refusal of Study Procedures or Unable to Take the Study Drug | 2 | 5 | 2
Not completed — Did Not Receive the Study Drug | 2 | 4 | 4

BASELINE CHARACTERISTICS:
Population: Baseline analysis population includes all randomized subjects who were administered at least one dose of study treatment (safety analysis set).
Groups:
- Total: Total of all reporting groups
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo | Total
Number analyzed (Participants) | 132 | 130 | 130 | 392
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (13.14) | 58.3 (13.07) | 58.5 (12.09) | 58.2 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 69 | 72 | 209
  Male | 64 | 61 | 58 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 13 | 27
  Not Hispanic or Latino | 125 | 121 | 116 | 362
  Unknown or Not Reported | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 1 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 6 | 10 | 29
  White | 109 | 118 | 110 | 337
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 4 | 4 | 7 | 15
BMI [Mean (Standard Deviation); unit: kg/m2] — Population: One subject in 7.5 g/day is excluded from the BMI calculation due to missing height.
  kg/m2
    number analyzed (Participants) | 132 | 129 | 130 | 391
    (all) | 28.43 (6.242) | 29.46 (5.788) | 28.97 (5.649) | 28.95 (5.900)

OUTCOME MEASURES:

1. Primary Outcome: Time to Gastrointestinal Recovery (GIR)
Description: Time to achieve recovery of GI motility as measured by a composite endpoint representing upper AND lower GI recovery
Time Frame: From the day after surgery (Day 1) until hospital discharge or Day 10 (whichever is earlier)
Population: Analysis population includes subjects in the Full Analysis Set in each treatment group who receive at least 1 dose of study medication, who underwent an elective bowel resection surgery as specified in the protocol, and who provided at least 1 post-surgery assessment of the primary endpoint (TGIR) during the treatment period.
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo
Number analyzed (Participants) | 132 | 128 | 130
hours | 32.6 [29.7 to 41.2] | 30.8 [28.1 to 35.3] | 33.4 [29.1 to 40.9]
Statistical Analysis 1: Comparison: TU-100 15 g/Day vs Placebo; Test type: Superiority; p = 0.767, Chi-squared — P-value is from the Wald Chi-Square statistic testing hypotheses of each dose of TU-100 compared with placebo: H0: hazard ratio (HR) = 1 vs. Ha: HR > 1; Cox Proportional Hazard = 0.91, 90% CI 2-sided [0.74 to 1.12] — Hazard ratio and confidence intervals (CIs) are derived from a Cox proportional hazard model that includes main effects for treatment and surgical approach
Statistical Analysis 2: Comparison: TU-100 7.5 g/Day vs Placebo; Test type: Superiority; p = 0.107, Chi-squared — P-value is from the Wald Chi-Square statistic testing hypotheses of each dose of TU-100 compared with placebo: H0: HR = 1 vs. Ha: HR > 1; Cox Proportional Hazard = 1.17, 90% CI 2-sided [0.95 to 1.44] — Hazard ratio and CIs are derived from a Cox proportional hazard model that includes main effects for treatment and surgical approach

2. Secondary Outcome: Time to GIR Responses
Description: Time to achieve first toleration of solid diet AND first bowel movement (Time to GI-2), time to first toleration of clear liquids, and time to absence of distension and presence of bowel sounds and flatus
Time Frame: From the day after surgery (Day 1) until hospital discharge or Day 10 (whichever is earlier)
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo
Number analyzed (Participants) | 132 | 128 | 130
hours
  Median Time to GI-2 | 49.4 [44.8 to 57.6] | 45.2 [43.5 to 46.8] | 47.2 [41.9 to 50.2]
  Median Time to first toleration of clear liquids | 24.0 [22.6 to 25.5] | 22.5 [21.2 to 23.6] | 23.3 [22.6 to 24.9]
  Median Time to absence of distension and presence of bowel sounds and flatus | 38.2 [31.3 to 41.8] | 40.1 [30.7 to 43.7] | 41.2 [37.8 to 44.6]
Statistical Analysis 1: Comparison: TU-100 15 g/Day vs Placebo; For Time to GI-2; Test type: Superiority; p = 0.780, Chi-squared — [p-value comment as in outcome 1, analysis 2]; Cox Proportional Hazard = 0.90, 90% CI 2-sided [0.71 to 1.13] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: TU-100 7.5 g/Day vs Placebo; For Time to GI-2; Test type: Superiority; p = 0.330, Chi-squared — [p-value comment as in outcome 1, analysis 2]; Cox Proportional Hazard = 1.06, 90% CI 2-sided [0.84 to 1.34] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: TU-100 15 g/Day vs Placebo; For Time to first toleration of clear liquids; Test type: Superiority; p = 0.788, Chi-squared — [p-value comment as in outcome 1, analysis 2]; Cox Proportional Hazard = 0.90, 90% CI 2-sided [0.73 to 1.11] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: TU-100 7.5 g/Day vs Placebo; For Time to first toleration of clear liquids; Test type: Superiority; p = 0.055, Chi-squared — [p-value comment as in outcome 1, analysis 2]; Cox Proportional Hazard = 1.22, 90% CI 2-sided [0.99 to 1.51] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: TU-100 15 g/Day vs Placebo; For Time to absence of distension and presence of bowel sounds and flatus; Test type: Superiority; p = 0.306, Chi-squared — [p-value comment as in outcome 1, analysis 2]; Cox Proportional Hazard = 1.07, 90% CI 2-sided [0.86 to 1.32] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: TU-100 7.5 g/Day vs Placebo; For Time to absence of distension and presence of bowel sounds and flatus; Test type: Superiority; p = 0.243, Chi-squared — [p-value comment as in outcome 1, analysis 2]; Cox Proportional Hazard = 1.09, 90% CI 2-sided [0.88 to 1.35] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Time to Discharge
Description: Time at which the subject is considered ready for discharge by the investigator based solely on GI recovery (Time to ready for discharge), and time at which the investigator writes discharge order for the subject (Time to discharge order written)
Time Frame: From surgery to hospital discharge
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo
Number analyzed (Participants) | 132 | 128 | 130
hours
  Time to ready for discharge | 56.1 [49.4 to 66.3] | 52.2 [48.4 to 59.8] | 66.1 [52.4 to 68.2]
  Time to discharge order written | 64.3 [50.5 to 67.8] | 58.1 [51.1 to 65.7] | 66.6 [63.5 to 69.1]
Statistical Analysis 1: Comparison: TU-100 15 g/Day vs Placebo; For Time to ready for discharge; Test type: Superiority; p = 0.489, Chi-squared — [p-value comment as in outcome 1, analysis 2]; Cox Proportional Hazard = 1.00, 90% CI 2-sided [0.81 to 1.24] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: TU-100 7.5 g/Day vs Placebo; For Time to ready for discharge; Test type: Superiority; p = 0.138, Chi-squared — [p-value comment as in outcome 1, analysis 2]; Cox Proportional Hazard = 1.15, 90% CI 2-sided [0.93 to 1.42] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: TU-100 15 g/Day vs Placebo; For Time to discharge order written; Test type: Superiority; p = 0.473, Chi-squared — [p-value comment as in outcome 1, analysis 2]; Cox Proportional Hazard = 1.01, 90% CI 2-sided [0.82 to 1.24] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: TU-100 7.5 g/Day vs Placebo; For Time to discharge order written; Test type: Superiority; p = 0.045, Chi-squared — [p-value comment as in outcome 1, analysis 2]; Cox Proportional Hazard = 1.24, 90% CI 2-sided [1.01 to 1.53] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: GIR Outcome Related to Length of Hospitalization (Mean)
Description: Mean number of days that the subject stayed in the hospital calculated based on calendar day of discharge order written
Time Frame: From surgery to hospital discharge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo
Number analyzed (Participants) | 132 | 128 | 130
days | 3.3 (3.07) | 2.7 (1.30) | 3.3 (3.00)
Statistical Analysis 1: Comparison: TU-100 15 g/Day vs Placebo; Test type: Superiority; p = 0.923, t-test, 2 sided — P-value is from two-sample t-test comparing TU-100 15 g/day treatment group versus placebo
Statistical Analysis 2: Comparison: TU-100 7.5 g/Day vs Placebo; Test type: Superiority; p = 0.039, t-test, 2 sided — P-value is from two-sample t-test comparing TU-100 7.5 g/day treatment group versus placebo

5. Secondary Outcome: GIR Outcome Related to Length of Hospitalization (Median)
Description: Median number of days that the subject stayed in the hospital calculated based on calendar day of discharge order written
Time Frame: From surgery to hospital discharge
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo
Number analyzed (Participants) | 132 | 128 | 130
days | 3 [1 to 28] | 2 [1 to 7] | 3 [1 to 29]

6. Secondary Outcome: Percentage of GIR Responders
Description: Percentage of subjects who achieve GIR (GIR responders) by day
Time Frame: From the day after surgery (Day 1) until hospital discharge or Day 10 (whichever is earlier)
Population: Analysis population includes subjects in the Full Analysis population in each treatment group who receive at least 1 dose of study medication, who underwent an elective BR surgery as specified in the protocol, and who provided at least 1 post-surgery assessment of the primary endpoint (TGIR) during the treatment period.
Measure: Number; unit: percentage of subjects
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo
Number analyzed (Participants) | 132 | 128 | 130
percentage of subjects
  Day 1 | 20.5 | 22.7 | 24.6
  Day 2 | 47.0 | 55.5 | 42.3
  Day 3 | 18.2 | 14.1 | 20.8
  Day 4 | 3.8 | 1.6 | 6.2
Statistical Analysis 1: Comparison: TU-100 15 g/Day vs Placebo; For Day 1; Test type: Superiority; p = 0.434, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.44 to 1.42] — Responder status is analyzed using logistic regression with GIR response as the dependent variable; treatment and surgical approach (open, laparoscopic) as covariates
Statistical Analysis 2: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 1; Test type: Superiority; p = 0.710, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.51 to 1.59] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: TU-100 15 g/Day vs Placebo; For Day 2; Test type: Superiority; p = 0.410, Chi-squared — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.75 to 2.02] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 2; Test type: Superiority; p = 0.037, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 1.70, 95% CI 2-sided [1.03 to 2.81] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: TU-100 15 g/Day vs Placebo; For Day 3; Test type: Superiority; p = 0.579, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.46 to 1.55] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 3; Test type: Superiority; p = 0.167, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.33 to 1.21]
Statistical Analysis 7: Comparison: TU-100 15 g/Day vs Placebo; For Day 4; Test type: Superiority; p = 0.400, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.21 to 1.86] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 4; Test type: Superiority; p = 0.083, Regression, Logistic; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.07 to 1.18] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: POI-related Morbidity
Description: Primary POI that is not secondary to surgical complication, such as anastomotic leak, abscess formation, or sepsis that requires readmission within 7 days of discharge, or need for postoperative nasal gastric tube insertion to manage symptoms of POI (vomiting/retching, abdominal distension)
Time Frame: From the day after surgery to discharge follow-up visit (30 days (+ 15 days) after hospital discharge)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo
Number analyzed (Participants) | 132 | 128 | 130
Participants | 7 | 5 | 5
Statistical Analysis 1: Comparison: TU-100 15 g/Day vs Placebo; Test type: Superiority; p = 0.621, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.43 to 4.14] — POI-related Morbidity status is analyzed using logistic regression with POI-related morbidity as the dependent variable; treatment and surgical approach (open, laparoscopic) as covariates
Statistical Analysis 2: Comparison: TU-100 7.5 g/Day vs Placebo; Test type: Superiority; p = 0.962, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.31 to 3.46] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of patients with adverse events (AEs) observed following administration of TU-100.
Time Frame: From baseline to discharge follow-up visit (30 days (+ 15 days) after hospital discharge)
Population: Analysis population includes all randomized subjects who were administered at least one dose of study treatment (safety analysis set). More details on patient incidence of adverse events (AEs) observed following administration of TU-100 is entered in AE section.
Measure: Count of Participants; unit: Participants
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo
Number analyzed (Participants) | 132 | 128 | 130
Participants | 78 | 73 | 81

9. Other Pre Specified Outcome: Subject-Reported Occurrence of Nausea
Description: Subjects will record the occurrence of nausea in their eDiaries on all postoperative in-hospital days.
Time Frame: From the day after surgery (Day 1) until hospital discharge or Day 10 (whichever is earlier)
Population: Analysis population includes subjects in the Full Analysis population in each treatment group who receive at least 1 dose of study medication, who underwent an elective BR surgery as specified in the protocol, and who answered to the questionnaire through the eDiaries. The questionnaire is only answered during hospital stays, and data is no longer collected once the subjects are discharged. Number Analyzed for each day represents number of subject answered the questionnaire for the day.
Measure: Count of Participants; unit: Participants
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo
Number analyzed (Participants) | 104 | 101 | 103
Participants
  Day 1 | 39 | 37 | 35
  Day 2: number analyzed (Participants) | 50 | 51 | 67
  Day 2 | 26 | 16 | 25
  Day 3: number analyzed (Participants) | 21 | 20 | 29
  Day 3 | 10 | 9 | 11
  Day 4: number analyzed (Participants) | 10 | 11 | 15
  Day 4 | 3 | 6 | 6
Statistical Analysis 1: Comparison: TU-100 15 g/Day vs Placebo; For Day 1; Test type: Superiority; p = 0.604, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.66 to 2.05] — Subject-reported (eDiary) - Nausea status is analyzed using logistic regression with Subject-reported (eDiary) - Nausea as the dependent variable; treatment and surgical approach (open, laparoscopic) as covariates
Statistical Analysis 2: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 1; Test type: Superiority; p = 0.693, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.63 to 1.99] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: TU-100 15 g/Day vs Placebo; For Day 2; Test type: Superiority; p = 0.122, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.85 to 3.78] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 2; Test type: Superiority; p = 0.518, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.36 to 1.67] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: TU-100 15 g/Day vs Placebo; For Day 3; Test type: Superiority; p = 0.528, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.46 to 4.53] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 3; Test type: Superiority; p = 0.689, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.40 to 4.07] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: TU-100 15 g/Day vs Placebo; For Day 4; Test type: Superiority; p = 0.653, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.12 to 3.70] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 8: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 4; Test type: Superiority; p = 0.452, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 1.85, 95% CI 2-sided [0.37 to 9.25] — [estimate comment as in outcome 9, analysis 1]

10. Other Pre Specified Outcome: Subject-Reported Bothersomeness of Nausea
Description: Subjects who answered that they felt nauseous will record bothersomeness of nausea in their eDiaries on all postoperative in-hospital days. Bothersomeness is measured on a scale of 0-10 with 10 being the most bothersome.
Time Frame: From the day after surgery (Day 1) until hospital discharge or Day 10 (whichever is earlier)
Population: Analysis population includes subjects in the Full Analysis population in each treatment group who receive at least 1 dose of study medication, who underwent an elective BR surgery as specified in the protocol, and who answered that they felt nausea on the day in the questionnaire through the eDiaries. Data is collected during hospital stays, and no longer collected once the subjects are discharged. Number Analyzed for each day represents number of subject with data for the day.
Measure: Least Squares Mean (Standard Error); unit: score of nausea bothersomeness
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo
Number analyzed (Participants) | 40 | 38 | 35
score of nausea bothersomeness
  Day 1 | 5.5 (0.46) | 6.0 (0.47) | 6.1 (0.48)
  Day 2: number analyzed (Participants) | 26 | 16 | 25
  Day 2 | 6.0 (0.53) | 4.7 (0.66) | 5.8 (0.54)
  Day 3: number analyzed (Participants) | 11 | 9 | 11
  Day 3 | 6.7 (0.78) | 5.5 (0.86) | 6.5 (0.79)
Statistical Analysis 1: Comparison: TU-100 15 g/Day vs Placebo; For Day 1, least square (LS) mean difference between placebo and TU-100 15 g/day. Mixed Model Repeated Measures approach was used to assess the bothersomeness of Nausea as the dependent variable and treatment group, surgical approach and treatment group by visit as covariates. An unstructured covariance structure is used to model the within-subject errors, shared across treatments; Test type: Superiority; p = 0.359, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.8 to 0.6]
Statistical Analysis 2: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 1, LS mean difference between placebo and TU-100 7.5 g/day. Mixed Model Repeated Measures approach was used to assess the bothersomeness of Nausea as the dependent variable and treatment group, surgical approach and treatment group by visit as covariates. An unstructured covariance structure is used to model the within-subject errors, shared across treatments; Test type: Superiority; p = 0.907, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.3 to 1.2]
Statistical Analysis 3: Comparison: TU-100 15 g/Day vs Placebo; For Day 2, LS mean difference between placebo and TU-100 15 g/day. Mixed Model Repeated Measures approach was used to assess the bothersomeness of Nausea as the dependent variable and treatment group, surgical approach and treatment group by visit as covariates. An unstructured covariance structure is used to model the within-subject errors, shared across treatments; Test type: Superiority; p = 0.856, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.3 to 1.6]
Statistical Analysis 4: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 2, LS mean difference between placebo and TU-100 7.5 g/day. Mixed Model Repeated Measures approach was used to assess the bothersomeness of Nausea as the dependent variable and treatment group, surgical approach and treatment group by visit as covariates. An unstructured covariance structure is used to model the within-subject errors, shared across treatments; Test type: Superiority; p = 0.180, Mixed Models Analysis; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.7 to 0.5]
Statistical Analysis 5: Comparison: TU-100 15 g/Day vs Placebo; For Day 3, LS mean difference between placebo and TU-100 15 g/day. Mixed Model Repeated Measures approach was used to assess the bothersomeness of Nausea as the dependent variable and treatment group, surgical approach and treatment group by visit as covariates. An unstructured covariance structure is used to model the within-subject errors, shared across treatments; Test type: Superiority; p = 0.814, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.9 to 2.4]
Statistical Analysis 6: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 3, LS mean difference between placebo and TU-100 7.5 g/day. Mixed Model Repeated Measures approach was used to assess the bothersomeness of Nausea as the dependent variable and treatment group, surgical approach and treatment group by visit as covariates. An unstructured covariance structure is used to model the within-subject errors, shared across treatments; Test type: Superiority; p = 0.409, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-3.2 to 1.3]

11. Other Pre Specified Outcome: Subject-Reported Occurrence of Abdominal Bloating
Description: Subjects will record the occurrence of abdominal bloating in their eDiaries on all postoperative in-hospital days.
Time Frame: From the day after surgery (Day 1) until hospital discharge or Day 10 (whichever is earlier)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo
Number analyzed (Participants) | 104 | 101 | 103
Participants
  Day 1 | 61 | 67 | 66
  Day 2: number analyzed (Participants) | 50 | 51 | 67
  Day 2 | 30 | 30 | 49
  Day 3: number analyzed (Participants) | 21 | 20 | 29
  Day 3 | 14 | 13 | 21
  Day 4: number analyzed (Participants) | 10 | 11 | 15
  Day 4 | 6 | 7 | 11
Statistical Analysis 1: Comparison: TU-100 15 g/Day vs Placebo; For Day 1; Test type: Superiority; p = 0.430, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.46 to 1.40] — Subject-reported (eDiary) - Abdominal Bloating status is analyzed using logistic regression with Subject-reported (eDiary) - Abdominal Bloating as the dependent variable; treatment and surgical approach (open, laparoscopic) as covariates
Statistical Analysis 2: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 1; Test type: Superiority; p = 0.739, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.62 to 1.96] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: TU-100 15 g/Day vs Placebo; For Day 2; Test type: Superiority; p = 0.130, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.25 to 1.20] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 2; Test type: Superiority; p = 0.099, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.24 to 1.13] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: TU-100 15 g/Day vs Placebo; For Day 3; Test type: Superiority; p = 0.686, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.23 to 2.63] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 3; Test type: Superiority; p = 0.644, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.22 to 2.56] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: TU-100 15 g/Day vs Placebo; For Day 4; Test type: Superiority; p = 0.498, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.09 to 3.18] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 4; Test type: Superiority; p = 0.700, Regression, Logistic — p value is assessing the null hypothesis that the odds ratio is equal to 1; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.12 to 4.05] — [estimate comment as in outcome 11, analysis 1]

12. Other Pre Specified Outcome: Subject-Reported Bothersomeness of Abdominal Bloating
Description: Subjects who answered that they felt bloated will record bothersomeness of abdominal bloating in their eDiaries on all postoperative in-hospital days. Bothersomeness is measured on a scale of 0-10 with 10 being the most bothersome.
Time Frame: From the day after surgery (Day 1) until hospital discharge or Day 10 (whichever is earlier)
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: score of bloating bothersomeness
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo
Number analyzed (Participants) | 62 | 67 | 66
score of bloating bothersomeness
  Day 1 | 5.2 (0.34) | 4.2 (0.33) | 5.2 (0.33)
  Day 2: number analyzed (Participants) | 30 | 30 | 49
  Day 2 | 5.6 (0.44) | 4.4 (0.43) | 4.6 (0.36)
  Day 3: number analyzed (Participants) | 14 | 13 | 21
  Day 3 | 5.6 (0.62) | 4.3 (0.64) | 5.0 (0.51)
Statistical Analysis 1: Comparison: TU-100 15 g/Day vs Placebo; For Day 1, LS mean difference between placebo and TU-100 15 g/day. Mixed Model Repeated Measures approach was used to assess the bothersomeness of Abdominal Bloating as the dependent variable and treatment group, surgical approach and treatment group by visit as covariates. An unstructured covariance structure is used to model the within-subject errors, shared across treatments; Test type: Superiority; p = 0.919, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.9 to 0.8]
Statistical Analysis 2: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 1, LS mean difference between placebo and TU-100 7.5 g/day. Mixed Model Repeated Measures approach was used to assess the bothersomeness of Abdominal Bloating as the dependent variable and treatment group, surgical approach and treatment group by visit as covariates. An unstructured covariance structure is used to model the within-subject errors, shared across treatments; Test type: Superiority; p = 0.016, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.8 to -0.2]
Statistical Analysis 3: Comparison: TU-100 15 g/Day vs Placebo; For Day 2, LS mean difference between placebo and TU-100 15 g/day. Mixed Model Repeated Measures approach was used to assess the bothersomeness of Abdominal Bloating as the dependent variable and treatment group, surgical approach and treatment group by visit as covariates. An unstructured covariance structure is used to model the within-subject errors, shared across treatments; Test type: Superiority; p = 0.064, Mixed Models Analysis; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-0.1 to 2.0]
Statistical Analysis 4: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 2, LS mean difference between placebo and TU-100 7.5 g/day. Mixed Model Repeated Measures approach was used to assess the bothersomeness of Abdominal Bloating as the dependent variable and treatment group, surgical approach and treatment group by visit as covariates. An unstructured covariance structure is used to model the within-subject errors, shared across treatments; Test type: Superiority; p = 0.683, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.3 to 0.8]
Statistical Analysis 5: Comparison: TU-100 15 g/Day vs Placebo; For Day 3, LS mean difference between placebo and TU-100 15 g/day. Mixed Model Repeated Measures approach was used to assess the bothersomeness of Abdominal Bloating as the dependent variable and treatment group, surgical approach and treatment group by visit as covariates. An unstructured covariance structure is used to model the within-subject errors, shared across treatments; Test type: Superiority; p = 0.462, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.0 to 2.1]
Statistical Analysis 6: Comparison: TU-100 7.5 g/Day vs Placebo; For Day 3, LS mean difference between placebo and TU-100 7.5 g/day. Mixed Model Repeated Measures approach was used to assess the bothersomeness of Abdominal Bloating as the dependent variable and treatment group, surgical approach and treatment group by visit as covariates. An unstructured covariance structure is used to model the within-subject errors, shared across treatments; Test type: Superiority; p = 0.343, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.3 to 0.8]

ADVERSE EVENTS:
Time Frame: From baseline to discharge follow-up visit (30 days (+ 15 days) after hospital discharge)
Description: Adverse Events reported in all randomized subjects who receive at least 1 dose of study drug.
Arm/Group | TU-100 15 g/Day | TU-100 7.5 g/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/130 | 0/130
Serious Adverse Events (participants affected / at risk) | 19/132 | 14/130 | 9/130
Other Adverse Events (participants affected / at risk) | 29/132 | 39/130 | 39/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TU-100 15 g/Day (N=132) | TU-100 7.5 g/Day (N=130) | Placebo (N=130)
Postoperative ileus (Injury, poisoning and procedural complications) | 8 | 3 | 3
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 2 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal mucosal tear (Gastrointestinal disorders) | 1 | 0 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TU-100 15 g/Day (N=132) | TU-100 7.5 g/Day (N=130) | Placebo (N=130)
Nausea (Gastrointestinal disorders) | 16 | 20 | 25
Vomiting (Gastrointestinal disorders) | 10 | 10 | 8
Abdominal distension (Gastrointestinal disorders) | 5 | 7 | 5
Constipation (Gastrointestinal disorders) | 2 | 8 | 7
Diarrhoea (Gastrointestinal disorders) | 7 | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT04742907/Prot_SAP_000.pdf